CLINICAL TRIAL: NCT07271485
Title: Randomized, Placebo-Controlled Pilot Study of Propranolol for Treating Misophonia
Brief Title: Propranolol for Misophonia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bloom Mental Health, LLC (Other)
Responsible Party: Principal Investigator, Jadon Webb, Principal Investigator, Bloom Mental Health, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 824
Record Dates: First submitted 2025-11-20; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Misophonia; Propanolol; Misophonia Treatment
MeSH Terms: conditions — misophonia | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propranolol Pill (Experimental): 10 participants will take one-time dose of 20 mg propranolol pill
  Interventions: Drug: propranolol
- Placebo Pill (Placebo Comparator): 10 participants will take be given a matching one-time dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: propranolol — A one-time dose of 20 mg propranolol
  Arms: Propranolol Pill
Drug: Placebo — A dose of placebo taken orally
  Arms: Placebo Pill

SUMMARY:
The primary goal of this study is to investigate whether a one-time dose of 20 mg oral propranolol can temporarily reduce the adverse emotional and physical symptoms triggered by misophonia.

The secondary goals of this study are:

1. Determine potential predictors of response to propranolol treatment, including demographic factors, baseline symptom severity, psychometric instrument item responses, and physiological characteristics.
2. Evaluate the safety and tolerability of propranolol in individuals with misophonia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Able to complete study visit(s) in Littleton, CO.
* Able to give informed consent.
* Participant reports clinically significant misophonia symptoms, as determined by answers on the standardized "Misophonia Trigger Screening Questions for Participants" form (described separately in the protocol). Specifically, participants must demonstrate relevant misophonia trigger responses that meet pre-specified minimum severity criteria detailed on this form.
* A-MISO-S rating scale severity criterion: Participants must score at least a moderate ("2") or higher on question 2 and question 3 of the Amsterdam Misophonia Scale (A-MISO-S) at screening, since this indicates clinically meaningful misophonia severity for study eligibility.
* Able to communicate misophonic distress in writing and reasonably participate in our outpatient clinical setting, meaning able to tolerate being in this outpatient clinical setting, follow the clinic rules for all patients and guests, and respond in an understandable fashion to questions administered to them.
* Must agree to follow study clinician advice and seek additional care outside of this clinic if advised (e.g., if advised to seek help from emergency services for a potentially serious adverse reaction).
* English fluency

Exclusion Criteria:

* Current use of scheduled propranolol for any condition.
* Any of the known contraindications for taking propranolol:
* cardiogenic shock
* sinus bradycardia (<50 bpm)
* greater than first degree heart block
* BP below 90/60
* asthma / bronchial asthma that requires treatment or medication, and/or has caused clinical concerns within the last 5 years
* Other heart conditions that require ongoing medical treatment
* Participants with any of the following relative contraindications for taking propranolol:
* participants who have active anorexia, purging, or who are underweight (<18.5 BMI)
* Active drug or alcohol use within the last 48 hours prior to study participation, or active drug withdrawals
* A history of untreated diabetes or other endocrine disorders that could be harmed by exposure to propranolol
* history of cardiovascular disease or stroke, or symptomatic blood disorders such as anemia
* history of any other severe physical or neurological conditions that may affect their ability to participate in the study
* Participants with liver or kidney disease that would be affect or be affected by the study drug
* Participants may, depending on the circumstances as decided by the study clinician, be excluded for any of the following conditions that may have adverse reactions to propranolol, including: Raynaud disease or other peripheral vascular disease, Pheochromocytoma, Psoriasis, Thyroid disease (untreated, and affected by propranolol), Unexplained dizziness, Oxygen level below 91%, Respirations below 12 or above 20
* Participants taking any other medications that could interfere with the effects of propranolol, as determined by the study clinician (e.g. other beta blockers, alpha blockers,prazosin, clonidine, guanfacine, diuretics, calcium channel blockers, acute us of anti-anxiety medications; other medications that interfere with the adrenergic system; or medications that have a significant effect on propranolol's pharmacology that would normally affect dosing in clinical practice
* Allergy or sensitivity to propranolol, placebo ingredients, and/or capsule ingredients.
* Pregnant or nursing.
* Any of the following in 30 days prior to enrollment: active psychosis, suicidal/ self-harming / homicidal thoughts, bipolar mania, panic attacks, traumatic dissociation, Post-Traumatic Stress Disorder (PTSD) flashbacks, or psychiatric hospitalization.
* Participant self-reports or clinical interview identifies any misophonia-triggered reactions within the past year that posed a significant risk to health or safety, including suicidal or homicidal ideation, or uncontrolled physical behaviors (e.g., self-injury, aggression toward others, throwing objects, screaming, or fleeing uncontrollably). This criterion is assessed via direct structured questioning during participant screening interviews and review of participant self-reports on standardized screening questionnaires.
* Misophonia trigger symptoms are determined by a medical provider to be better explained by a condition other than Misophonia, such as hyperacusis or phonophobia.
* Inability to hear routine sounds and communication (ie severe hearing impairment), only if it interferes with ability to hear the misophonia triggers on the video.
* Participants who are triggered by the sound of water running or a car alarm (our control videos)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Heart rate is continuously monitored via pulse oximetry during each video presentation. The continuous measurement will start at pre-intervention and end after the intervention.
  Heart rate was chosen as a primary biometric outcome because it reliably indicates sympathetic nervous system activation commonly observed in acute misophonia reactions. Given propranolol's established pharmacologic effect as a beta-blocker, the hypothesis is that propranolol will significantly blunt the heart rate increase typically elicited by misophonia triggers compared to placebo.
Visual Analog Scale (VAS) | The scale will be taken immediately after each video clip intervention. It will measure the participant's reaction to each clip.
  The Visual Analog Scale (VAS) assesses three core emotional domains (anger, anxiety, disgust) and multiple physical sensations frequently reported during acute misophonia episodes, such as feeling hot/sweaty, heart pounding, muscle tension, trembling/shaking, and shortness of breath. Each response is rated on a sliding scale accompanied by emojis or graphics that visually represent increasing intensity of the sensations or emotions. This format leverages established evidence from acute pain and emotional-response research, demonstrating that visual analogue scales effectively capture immediate subjective states. The VAS is based on a Likert scales ranging from 0-7, 0-5, and 0-8 in some questions. Higher scores indicates more distress and a worst outcome.

SECONDARY OUTCOMES:
Grip Strength | Grip Strength measurement is subsequently performed immediately after each video exposure. This will be taken immediately after each video clip intervention in order to measure the participant's reaction to each clip.
  An innovative exploratory measure of emotional and physical intensity will also be collected using a Grip Strength Meter. This measure is specifically designed for this study to provide participants with a physical, embodied way to express their subjective feelings of anger, distress, or tension following trigger exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- Bloom Mental Health, Littleton, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided